CLINICAL TRIAL: NCT00100906
Title: Randomized Phase II Trial Of Sequential ATRA Then IL-2 For Modulation Of Dendritic Cells And Treatment Of Metastatic Renal Cancer
Brief Title: Sequential ATRA Then IL-2 for Modulation of Dendritic Cells and Treatment of Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH); Chiron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13920; CA101324 (Other Grant/Funding Number: NIH); CA84488 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-07

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; clear cell renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Interleukin-2; aldesleukin; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ATRA Followed by IL-2 - Dose Level A (Active Comparator): Patients were assigned to one of three ATRA dose levels, at a 1:1:1 ratio, using a randomly permuted list assignments, with the assignment generally being made on the initial day of treatment.
  Week 1: One dose daily of IL-2 for 5 days followed by 2 days off.
  Weeks 2-6: One dose daily of IL-2 for 5 days followed by 2 days off.
  After the IL-2: 2-3 weeks rest, with no treatment. During this time a repeat physical exam, history and X-ray scans will be performed. If there has not been progression (worsening) of the patient's tumor, they will continue to a second 8-week treatment schedule.
  This schedule will be the same as the first, unless the patients dose had to be reduced. If so, patient's will get that reduced dose. It consists of 1 week of ATRA, 1 week of rest, followed by 6 weeks of IL-2. The same blood tests are collected during that second cycle.
  Interventions: Drug: IL-2; Drug: ATRA
- ATRA Followed by IL-2 - Dose Level B (Active Comparator): Patients were assigned to one of three ATRA dose levels, at a 1:1:1 ratio, using a randomly permuted list assignments, with the assignment generally being made on the initial day of treatment.
  Week 1: One dose daily of IL-2 for 5 days followed by 2 days off.
  Weeks 2-6: One dose daily of IL-2 for 5 days followed by 2 days off.
  After the IL-2: 2-3 weeks rest, with no treatment. During this time a repeat physical exam, history and X-ray scans will be performed. If there has not been progression (worsening) of the patient's tumor, they will continue to a second 8-week treatment schedule.
  This schedule will be the same as the first, unless the patients dose had to be reduced. If so, patient's will get that reduced dose. It consists of 1 week of ATRA, 1 week of rest, followed by 6 weeks of IL-2. The same blood tests are collected during that second cycle.
  Interventions: Drug: IL-2; Drug: ATRA
- ATRA Followed by IL-2 - Level C (Active Comparator): Patients were assigned to one of three ATRA dose levels, at a 1:1:1 ratio, using a randomly permuted list assignments, with the assignment generally being made on the initial day of treatment.
  Week 1: One dose daily of IL-2 for 5 days followed by 2 days off.
  Weeks 2-6: One dose daily of IL-2 for 5 days followed by 2 days off.
  After the IL-2: 2-3 weeks rest, with no treatment. During this time a repeat physical exam, history and X-ray scans will be performed. If there has not been progression (worsening) of the patient's tumor, they will continue to a second 8-week treatment schedule.
  This schedule will be the same as the first, unless the patients dose had to be reduced. If so, patient's will get that reduced dose. It consists of 1 week of ATRA, 1 week of rest, followed by 6 weeks of IL-2. The same blood tests are collected during that second cycle.
  Interventions: Drug: IL-2; Drug: ATRA

INTERVENTIONS:
Drug: IL-2 — Immunotherapy with interleukin-2
  Other Names: interleukin-2; aldesleukin; Proleukin™; Recombinant Human Interleukin-2
Drug: ATRA
  Other Names: tretinoin; Vesanoid™; all-trans retinoic acid

SUMMARY:
RATIONALE: Tretinoin may help cells that are involved in the body's immune response to work better. Interleukin-2 may stimulate the white blood cells to kill kidney cancer cells. Giving tretinoin together with interleukin-2 may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well giving three different doses of tretinoin together with interleukin-2 works in treating patients with stage IV kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the ratio of dendritic cells (DC) to circulating immature cells (ImC) before and after treatment with 3 different doses of tretinoin in patients with stage IV renal cell cancer.
* Assess in vitro immune response assays to tetanus toxoid and influenza virus peptide before and after treatment with tretinoin and interleukin-2 in these patients.

Secondary

* Determine the frequency of treatment-related side effects in these patients.
* Determine clinical objective response and progression-free survival of patients treated with this regimen.
* Correlate DC:ImC ratio with clinical objective response in patients treated with this regimen.
* Correlate the extent of change of the DC:ImC ratio with tretinoin dose and tretinoin blood levels in these patients.

OUTLINE: This is a randomized, open-label study. Specimens are stratified according to patient prognostic factors, tumor bulk, and extent of dendritic cell to circulating immature cell ratio derangement. Patients are randomized to 1 of 3 tretinoin doses.

Patients are followed for up to 2 years.

PROJECTED ACCRUAL: A total of 27-36 patients (9-12 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal cell cancer

  * Stage IV disease
  * Histology with clear cell component
* Metastatic OR incompletely resected disease
* Non-measurable disease allowed
* Underwent complete or partial nephrectomy more than 90 days ago

  * No unresected primary cancer
* No more than 2 of the following adverse factors:

  * Hemoglobin < 10.0 g/dL
  * Corrected calcium > upper limit of normal (ULN)
  * Lactic dehydrogenase > 1.5 times ULN
  * Eastern Cooperative Oncology Group (ECOG) performance status 2
* Brain metastasis allowed provided more than 90 days of clinical and radiologic stability after the end of its active treatment

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* See Disease Characteristics
* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* See Disease Characteristics
* Serum glutamic oxaloacetic transaminase (SGOT) < 3 times normal
* Bilirubin < 2 times normal

Renal

* See Disease Characteristics
* Creatinine clearance > 40 mL/min

Cardiovascular

* None of the following cardiovascular conditions within the past year:

  * Uncontrolled hypertension
  * Myocardial infarction
  * Unstable angina
  * New York Heart Association class II-IV congestive heart failure
  * Serious cardiac arrhythmia requiring medication
  * Class II-IV peripheral vascular disease within the past year
  * Other clinically significant cardiovascular disease

Immunologic

* No history of immunodeficiency disease
* No HIV infection
* No ongoing serious infection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use two methods of effective contraception during and for 1 month (for women) or 6 months (for men) after study treatment
* Other prior malignancy allowed provided there is no evidence of active disease
* No other medical contraindication to tretinoin or interleukin-2
* No serious non-healing wound, ulcer, or bone fracture

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 60 days since prior immunotherapy

Chemotherapy

* At least 60 days since prior cytotoxic chemotherapy

Endocrine therapy

* See Radiotherapy
* No prior corticosteroids at > physiologic replacement doses for > 3 days within the past 90 days
* Concurrent tamoxifen, toremifene, megestrol, or gonadotropin-releasing hormone agonists allowed
* Concurrent inhaled steroids allowed

Radiotherapy

* More than 7 days since prior external-beam radiotherapy

  * No steroid requirement during radiotherapy

Surgery

* See Disease Characteristics
* At least 30 days since other prior debulking surgery

Other

* Prior adjuvant therapy for resected, synchronous stage IV disease allowed
* Prior adjuvant therapy allowed

  * Study therapy is not to be used as adjuvant therapy for completely resected late (> 1 year until identification) solitary site of disease metastasis or non-metastatic disease
* No prior participation in this clinical study
* At least 60 days since other prior anticancer drugs
* Concurrent seizure medication allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-08; Primary Completion 2006-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Ratio of Dendritic Cells (DC) to Circulating Immature Cells (ImC) Before and After Treatment | 1 year, 3 months
  Determine the ratio of dendritic cells (DC) to circulating immature cells (ImC) before and after treatment with 3 different doses of tretinoin in patients with stage IV renal cell cancer.

SECONDARY OUTCOMES:
Frequency of Treatment-Related Side Effects | 1 year, 3 months
  Review of adverse events utilizing Common Toxicity Criteria (CTC) V3.
Overall Response Rate (ORR) | 1 year, 3 months
  Objective Response Rate according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Evaluate per-patient observed best clinical responses, after 11-12 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mayer Fishman, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- [Result] Mirza N, Fishman M, Fricke I, Dunn M, Neuger AM, Frost TJ, Lush RM, Antonia S, Gabrilovich DI. All-trans-retinoic acid improves differentiation of myeloid cells and immune response in cancer patients. Cancer Res. 2006 Sep 15;66(18):9299-307. doi: 10.1158/0008-5472.CAN-06-1690. PMID 16982775